CLINICAL TRIAL: NCT01506713
Title: Randomized, Open-label, 2-Way Crossover, Bioequivalence Study of Clopidogrel 75 mg Tablet With Plavix® 75 mg In Healthy Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Clopidogrel Tablets 75 mg of Dr. Reddy's Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 60280
Record Dates: First submitted 2012-01-06; First posted 2012-01-10 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Fasting
MeSH Terms: conditions — Fasting | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clopidogrel (Experimental): Clopidogrel tablets 75 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Clopidogrel
- Plavix (Active Comparator): Clopidogrel Tablet 75 mg
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel Tablets 75 mg
  Other Names: Plavix

SUMMARY:
The objective of this study was to compare the rate and extent of absorption of Dr. Reddy's Laboratories Ltd, clopidogrel and Bristol-Myers Squibb Company, USA Plavix®, clopidogrel 75 mg tablet under fasting condition.

DETAILED DESCRIPTION:
Randomized, Open-label, 2-Way Crossover, Bioequivalence Study of Clopidogrel 75 mg Tablet (Dr. Reddy's Laboratories Ltd., India) and Plavix® (Bristol-Myers Squibb Company, USA) Following a 75 mg Dose In Healthy Subjects Under Fasting Conditions.

ELIGIBILITY:
Inclusion Criteria:

Subjects enrolled in this study will be members of the community at large. The recruitment advertisements may use various media types (e.g. radio, newspaper, Anapharm Web site, Anapharm volunteers' database). Subjects must meet all of the following criteria to be included in the study:

* Male or female, non-smoker, ≥18 and ≤55 years of age.
* Medically healthy with clinically normal laboratory profile, vital signs and ECG.
* Capable of consent.
* BMI ≥19.0 and <30.0

Exclusion Criteria:

Subjects to whom any of the following applies will be excluded from the study:

* Clinically significant illness or surgery within 4 weeks prior to dosing.
* Any clinically significant abnormality or abnormal laboratory test results found during medical screening.
* Any reason which, in the opinion of the Clinical Sub-.investigator, would prevent the subject from participating in the study.
* Positive test for hepatitis B, hepatitis C, or HIV at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or• heart rate less than 50 or over J00 bpm) at screening.
* History of significant alcohol abuse or drug abuse within one year prior to the screening visit.
* Regular use of alcohol within six months prior to the screening visit (more than fourteen units of alcohol per week [J Unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]), or positive alcohol breath test at screening.
* Use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine (PCP] and -crack) within 1 year prior to the screening visit or positive urine drug screen at screening.
* History of allergic reactions to clopidogrel or other related drugs.
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; examples of inhibitors: antidepressants (SSRI), cimetidine, diltiazem, macrolides, imidazoles, neuroleptics, verapamil, fIuoroquinolones, antihistamines) within 30 days prior to administration of the study medication.
* Use of an investigational drug or participation in an investigational study within 30 days prior to dosing.
* Clinically significant history or presence of any gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug.
* Any clinically significant history or presence of neurological, endocrinal, cardiovascular, pulmonary, hematological, immunologic, psychiatric, or metabolic disease.
* Use of prescription medication within 14 days prior to administration of study medication or over-the counter products (including natural food supplements, vitamins, garlic as a supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption and hormonal contraceptives.
* Difficulty to swallow study medication.
* Use of any tobacco products in the 3 months preceding drug administration.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the Clinical Sub-Investigator, could contraindicate the subject's participation in this study.
* A depot injection or an implant of any drug (other than hormonal contraceptives) within 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 7 days prior to drug administration. Donation or loss of whole blood (excluding the volume of blood that will be drawn during the screening procedures of this study) prior to administration of the study medication as follows:
* 50 mL to 499 mL of whole blood within 30 days,
* more than 499 mL of whole blood within 56 days prior to drug administration.
* Positive urine pregnancy test at screening.
* Breast-feeding subject.
* Female subjects of childbearing potential having unprotected sexual intercourse with any non-sterile male partner (i.e. male who has not been sterilized by vasectomy for at least 6 months) within 14 days prior to study drug administration. Acceptable methods of contraception are:
* intra-uterine contraceptive device (placed at least 4 weeks prior to study drug administration;
* condom or diaphragm + spermicide;
* hormonal contraceptives (starting at least 4 weeks prior to study drug administration).
* History or known active pathological bleeding (e.g. peptic ulcer, intracranial hemorrhage).
* Increased risks of bleeding (e.g. frequent nose bleeding, recent trauma, surgery or other pathological condition).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2006-09; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Bioequivalence is based on Cmax and AUC parameters | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Denis Audet, MD, Principal Investigator — Anapharm
Locations (1):
- Anapharm, Sainte-Foy (Quebec), Canada